CLINICAL TRIAL: NCT03501784
Title: Nobio Antimicrobial Particles Effect in a Split Mouth Model
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nobio Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ND01 version 02
Record Dates: First submitted 2018-03-06; First posted 2018-04-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2018-08

CONDITIONS: Cervical Caries
MeSH Terms: conditions — Root Caries | interventions — Equipment and Supplies

STUDY DESIGN:
Intervention Model Description: This is an exploratory, comparative, self-controlled, single blind study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Novidia Dental bonding and flow (Experimental): Nobio particles incorporated within Novidia Dental Bonding and Flow.
  Interventions: Device: Nobio particles incorporated within Novidia Dental Bonding
- Filtek bond and flow composite (Active Comparator): standard of care class V composite restoration performed with Filtek and 3M
  Interventions: Device: Filtek bond and flow composite

INTERVENTIONS:
Device: Nobio particles incorporated within Novidia Dental Bonding — Nobio particles incorporated within Novidia Dental Bonding and Flow
  Other Names: Device
  Arms: Novidia Dental bonding and flow
Device: Filtek bond and flow composite — standard of care class V composite restoration performed with Filtek and 3M
  Arms: Filtek bond and flow composite

SUMMARY:
The study purpose is to evaluate the antimicrobial effect of Nobio particles incorporated within Novidia Dental Bonding and Flowable Composite versus standard of care within a split mouth model.The study population will include 35 subjects considered to be at high risk for cervical caries and affected by uncontrolled plaque accumulation

DETAILED DESCRIPTION:
An exploratory, comparative, self-controlled single blinded interventional study. Intended to evaluate the antimicrobial effect of Nobio particles incorporated within Novidia Dental Bonding and Flowable composite versus Filtek bond and flow composite within a split mouth model.The study population (N=35) will be high risk population for cervical caries (with at least 2 carious cavities in the mouth) affected by uncontrolled plaque accumulation.Each subject will serve in this model as his own control.On one side the Novidia intervention will be made and on the contralateral side the Filtek intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years of age.
* Requires two cervical restorations or the exchange of existing ones
* Subject has poor oral hygiene and at high risk for plaque accumulation.
* Subject able and willing to comply with study visits and Follow up visits and signed the informed consent.

Exclusion Criteria:

* Allergic reaction to iodide.
* Pregnant or lactating women.
* Use of antiseptic mouth rinse or antibiotic up to 2 weeks before the beginning of study.

Exclusion criteria for the chosen teeth for the study:

* Tooth designated for extraction in the following 6 month.
* Tooth designated to have a root canal treatment.
* Tooth or several teeth designated for periodontal surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2018-09-22 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence and severity of adverse events related to dental care | one year
  Record unanticipated adverse device-related events (UADE),Incidence and nature of serious adverse events (SAE).
  Incidence and nature of adverse events

SECONDARY OUTCOMES:
Plaque index rate | one year
  0 -No Plaque up to 3-Abundance plaque
Replica method for bacterial count | one year
  Impression matrix sampling the tooth bio film layer
Physician assessment of cervical restoration integrity | one year
  Marginal integrity of the performed restoration
Subject and Dentist satisfaction questionnaire | one year
  satisfaction questionnaire ranging from 1(strongly disagree )to 10 (strongly agree)
Dead/Live Staining of biofilm (Cyto 9) | one year
  CSLM quantitative measurement

CONTACTS AND LOCATIONS:
Overall Officials: Bertrude LEV DOR, DMD, Principal Investigator — MACCABIDENT ASSUTA; Bat sheva Levy, Study Director — Nobio Ltd.
Locations (1):
- Assuta Medical Center -Maccabident, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
The final study results will be shared

REFERENCES:
- [Background] Atar-Froyman L, Sharon A, Weiss EI, Houri-Haddad Y, Kesler-Shvero D, Domb AJ, Pilo R, Beyth N. Anti-biofilm properties of wound dressing incorporating nonrelease polycationic antimicrobials. Biomaterials. 2015 Apr;46:141-8. doi: 10.1016/j.biomaterials.2014.12.047. Epub 2015 Jan 28. PMID 25678123
- [Result] Beyth N, Yudovin-Farber I, Perez-Davidi M, Domb AJ, Weiss EI. Polyethyleneimine nanoparticles incorporated into resin composite cause cell death and trigger biofilm stress in vivo. Proc Natl Acad Sci U S A. 2010 Dec 21;107(51):22038-43. doi: 10.1073/pnas.1010341107. Epub 2010 Dec 3. PMID 21131569